CLINICAL TRIAL: NCT07378176
Title: Prognosis of Primary Aldosteronism: A Prospective Cohort Study
Acronym: PA-PROG
Status: Recruiting | Type: Observational
Sponsor: Xinjiang Medical University (Other)
Collaborators: First Affiliated Hospital of Chengdu Medical College (Other); First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Xiang Xie, Professor, Xinjiang Medical University
Other Study IDs: K202512-38
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Primary Aldosteronism
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary Aldosteronism Group: Screened, confirmed and subtyped according to the guidelines.

SUMMARY:
Primary aldosteronism (PA) is the most common cause of secondary hypertension, and patients with PA have a significantly higher risk of developing cardiovascular and renal complications compared with those with essential hypertension. However, PA remains substantially underdiagnosed and undertreated in clinical practice, and relevant research data on the short-term and long-term prognosis of PA patients in the Chinese population are particularly scarce. This is a multicenter, prospective cohort study designed to systematically collect real-world clinical data of PA patients, including baseline clinical characteristics, etiological subtypes, diagnostic and therapeutic strategies, and long-term follow-up outcomes. Through 5 years of standardized follow-up, this study will analyze the differences in treatment efficacy among PA patients with different pathological subtypes (e.g., adrenal adenoma, adrenal hyperplasia), evaluate the short-term therapeutic efficacy and long-term prognosis of PA patients undergoing different treatment modalities including pharmacotherapy, surgery and interventional therapy, and explore the risk factors for adverse clinical outcomes. Ultimately, it will provide high-quality real-world evidence-based data to optimize the clinical diagnosis and management of PA and improve the long-term prognosis of affected patients.

DETAILED DESCRIPTION:
This study conducts long-term follow-up observations on patients with primary aldosteronism (PA), dynamically tracks changes in their condition, and systematically collects information related to treatment regimens and health outcomes, aiming to ultimately achieve the following research objectives: clarify the proportion and regularity of PA patients achieving normalization of both blood pressure and relevant hormonal levels after treatment (i.e., the status of "complete cure"); analyze differences in therapeutic efficacy among PA patients with different pathological subtypes such as adrenal adenoma and adrenal hyperplasia; evaluate the impact of different treatment modalities including pharmacotherapy, surgery and interventional therapy on patients' long-term health; observe the trajectory changes of PA-induced damage to the heart, kidneys and blood vessels, as well as metabolic and cognitive function abnormalities; and screen for key factors influencing patients' blood pressure control efficacy and the occurrence of cardiovascular and cerebrovascular events.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 80 years old.
2. Biochemically confirmed diagnosis of Primary Aldosteronism (PA) according to contemporary guidelines (e.g., confirmed positive case detection test and confirmatory test).
3. Voluntary to sign the informed consent.

Exclusion Criteria:

1. patients with severe cardiac, hepatic or renal dysfunction;
2. Diagnosis of secondary hypertension other than PA.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of primary aldosteronism (PA) confirmed in accordance with current clinical guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of Major Adverse Cardiovascular Events (MACE) | From study enrollment until the end of the 60-month follow-up period.
  The proportion of patients who experience an adjudicated Major Adverse Cardiovascular Event (MACE), defined as a composite endpoint consisting of non-fatal myocardial infarction, non-fatal stroke, hospitalization for heart failure, or cardiovascular death.

SECONDARY OUTCOMES:
All-cause mortality | From study enrollment until the end of the 60-month follow-up period.
  Record of deaths from any cause during follow-up. Confirmed by medical records, family follow-up, or national death registration systems.
Blood pressure control rate | 12, 24, 36, 48, and 60 months.
  Proportion of participants achieving target office blood pressure at each visit. Target is defined as seated systolic BP < 140 mmHg and diastolic BP < 90 mmHg. For participants with diabetes mellitus or chronic kidney disease, the target is seated systolic BP < 130 mmHg and diastolic BP < 80 mmHg.
Incidence of new-onset atrial fibrillation (AF) | From study enrollment until the end of the 60-month follow-up period. Routine screening ECGs will be performed at 12, 24, 36, 48, and 60 months.
  The proportion of participants newly diagnosed with atrial fibrillation. Diagnosis requires confirmation by 12-lead electrocardiogram or at least 30 seconds of AF on a 24-hour Holter monitor, as documented in medical records.
Incidence of cognitive impairment(Mild Cognitive Impairment or dementia) | 12, 24, 36, 48, and 60 months.
  Proportion of participants with Mild Cognitive Impairment（MCI） or all-cause dementia at follow-up visits..
Plasma Aldosterone Concentration (PAC) | Baseline, 12, 24, 36, 48, and 60 months.
Plasma Renin Concentration (PRC) | Baseline, 12, 24, 36, 48, and 60 months.
Serum Potassium (K+) Level | Baseline, 12, 24, 36, 48, and 60 months.
Estimated Glomerular Filtration Rate (eGFR) | Baseline, 12, 24, 36, 48, and 60 months.
Urinary Albumin-to-Creatinine Ratio (UACR) | Baseline, 12, 24, 36, 48, and 60 months.
Left Ventricular Mass Index (LVMI) | Baseline, 12, 24, 36, 48, and 60 months.
Carotid Intima-Media Thickness (CIMT) | Baseline, 12, 24, 36, 48, and 60 months.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Xie, PhD, Study Chair — First Affiliated Hospital of Xinjiang Medical University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Chengdu Medical College, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No